CLINICAL TRIAL: NCT01344460
Title: Multicenter, Open-label Study to Evaluate the Safety and Efficacy (by Blinded Reading) of Gadobutrol-enhanced Magnetic Resonance Angiography (MRA) After a Single Injection of 0.1 mmol/kg of Gadobutrol in Subjects With Known or Suspected Renal Artery Disease
Brief Title: Gadobutrol Enhanced MRA of the Renal Arteries
Acronym: GRAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91759; 2010-023002-13 (EudraCT Number)
Record Dates: First submitted 2011-04-05; First posted 2011-04-29 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Renal Artery Obstruction
Keywords: magnetic resonance angiography (MRA) of the renal arteries
MeSH Terms: conditions — Renal Artery Obstruction | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — a single bolus injection of approx. 0.1mmol/kg

SUMMARY:
Subjects referred for a routine CTA (computed tomography angiography) or MRA (magnetic resonance angiography) will be invited to participate in the study and subjects will be involved in the study for between 2 and 12 days. Two to three visits to the study doctor will be required.

This study will compare the diagnostic results of Gadobutrol enhanced MRA images with MRA images taken without contrast agent using images from a CTA as the standard of reference, which may have been performed up to 60 days prior to enrolment. If a CTA has not been performed in this prior time period, a CTA is required for the study.

MRA and CTA images will be collected for an independent review (blinded read).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged ≥ 18 years
* Known or suspected renal artery disease based on any of the following:

  * Referred for evaluation of the renal arteries for clinically significant stenosis
  * Follow-up for a metallic stent in a renal artery
  * Prior imaging study (CTA) showing ≥ 50% renal artery stenosis (within 60 days prior to consent)
* Willingness to undergo the routine Contrast Enhanced Magnetic Resonance Angiography (CE MRA) examinations with gadobutrol.
* Willingness and ability to follow directions and complete all study procedures specified in the protocol.
* Females of childbearing potential only: Negative pregnancy test on the day of the MRA prior to administration of study drug.
* Written informed consent (IC), including information about the provisions of the Health Insurance Portability and Accountability Act (HIPAA) as applicable.

Exclusion Criteria:

* Pregnant or nursing (including pumping for storage and feeding)
* Received any other investigational product or participation in any other clinical trial within 30 days before enrollment into this study
* Previous enrolment into this study or into any other Bayer sponsored study using gadobutrol
* Contraindication to the MRA examinations (e.g. inability to hold breath; severe arrhythmias; very low cardiac output, severe claustrophobia, defibrillators or other metallic devices not approved for MRI)
* Contraindication to the use of Gd-containing contrast agents (including subjects with suspicion for or known to have Nefrogenic Systemic Fibrosis (NSF)
* History of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents
* Received any contrast agent within 72 hours before the study MRA, or scheduled receipt of any contrast agent within 24 hours after the study MRA (Note: This applies also to a CTA potentially scheduled during the course of the study.)
* Estimated glomerular filtration rate (eGFR) value < 30 ml/min/1.73 m2 derived from a serum creatinine result within 2 weeks before the gadobutrol injection. Any subject on hemodialysis or peritoneal dialysis is excluded from participation. Use the value obtained prior to and closest to the time of the MRA, if there are multiple creatinine values. (Do not use the core lab value if not available prior to the MRA.)
* Acute renal insufficiency of any intensity, either due to hepato-renal syndrome or occurring in the peri-operative liver transplantation period
* Severe cardiovascular disease (e.g. acute myocardial infarction [< 14 days], unstable angina, congestive heart failure New York Heart Association class IV) or known long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (59):
- United States (14):
  - Tucson, Arizona
  - Los Angeles, California
  - Orange, California
  - Jacksonville, Florida
  - Miami, Florida
  - Savannah, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Durham, North Carolina
  - Providence, Rhode Island
  - Memphis, Tennessee
  - San Antonio, Texas
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (3):
  - Adrogué, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Austria (3):
  - Innsbruck, Tyrol
  - Vienna
  - Wiener Neustadt
- Brazil (3):
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Colombia (4):
  - Medellín, Antioquia
  - Barranquilla, Atlántico
  - Cali, Valle del Cauca Department
  - Bogotá
- Czechia (4):
  - Brno
  - Olomouc
  - Pilsen
  - Prague
- France (4):
  - La Tronche
  - Paris
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (7):
  - Karlsruhe, Baden-Wurttemberg
  - Frankfurt am Main, Hesse
  - Münster, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
  - Jena, Thuringia
- Poland (4):
  - Krakow
  - Lodz
  - Lublin
  - Warsaw
- South Korea (3):
  - Seoul, Seoul Teugbyeolsi
  - Seoul
  - Suwon
- Switzerland (4):
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Olten, Canton of Solothurn
  - Zurich, Canton of Zurich
- Taiwan (4):
  - Taipei, Taipei
  - Kaoshiung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 study centers in 13 countries, between 16 May 2011 (first participant first visit) and 06 July 2012 (last participant last visit).
Pre-assignment Details: A total of 338 participants were screened, of which 317 were enrolled and 315 received the study drug. The 23 participants who did not receive the study drug included 9 screen failures and 12 premature discontinuations (10 participants withdrew consent and 2 participants for other reasons) and 2 participants never received the study drug.
Groups:
- Gadobutrol (Gadavist, BAY 86-4875): Gadobutrol was administered to all participants receiving study drug at the standard dose of 0.1 mmol/kg body weight (bw) by single intravenous (i.v.) bolus injection. During the course of the study, non-contrast magnetic resonance angiography (MRA) images were obtained before the administration of gadobutrol, and gadobutrol-enhanced MRA images were obtained after injection.
Period: Overall Study
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Started | 315 (Participants received study drug; Safety analysis set)
Fulfilled Requirements of FAS Population | 292 (Full analysis set (FAS))
Completed | 312
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Number analyzed (Participants) | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (16.9)
Age, Customized [Number; unit: participants]
  < 45 years | 92
  45 - 64 years | 111
  >= 65 years | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145
  Male | 170
Baseline Weight [Mean (Standard Deviation); unit: kilogram(s)] | 77.5 (16.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Assessable Vascular Segments Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Each vascular segment was visualized using unenhanced MRA and gadobutrol-enhanced MRA, characterized by the on-site investigators, three independent blinded readers (reader 1, 2 and 3) and majority readers (the outcome determined by at least two of the blinded readers). The segments were predefined to standardize the blinded reader evaluations. A segment was assessable if it was visualized along its entire length and if any region of stenosis, was measured reliably. There were 6 segments assessed per participant (3 segments in the right renal artery and 3 segments in the left renal artery) and up to 9 segments in participants with renal transplant.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category for both groups.
Measure: Number; unit: Percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
Number analyzed (segments) | 1764 | 1764
Percentage of segments
  Majority reader (n=292/1752) | 95.9 | 77.6
  Blinded reader 1 (n=292/1746) | 98.1 | 81.7
  Blinded reader 2 (n=292/1752) | 95.5 | 71.5
  Blinded reader 3 (n=292/1734) | 95.5 | 78.1
  Clinical investigators (n=292/1764) | 94.4 | 68.9
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Majority reader; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.000, McNemar; Cluster adjusted McNemar; Percentage difference = 18.3, 95% CI 2-sided [lower limit 15.2] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 1; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.000, McNemar; Cluster adjusted McNemar; Percentage difference = 16.4, 95% CI 2-sided [lower limit 13.2] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 2; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.000, McNemar; Cluster adjusted McNemar; Percentage difference = 24.0, 95% CI 2-sided [lower limit 20.5] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 3; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.000, McNemar; Percentage difference = 17.4, 95% CI 2-sided [lower limit 14.3] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Clinical investigator; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.000, McNemar; Percentage difference = 25.6, 95% CI 2-sided [lower limit 21.9] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

2. Primary Outcome: Sensitivity for Detection of Clinically Significant Disease Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Clinically significant disease was defined as 50 to 99 percent (%) stenosis of a segment, but not occluded as assessed by the SoR. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of sensitivity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 113 | 113
Number analyzed (segments) | 140 | 140
percentage of sensitivity
  Majority reader | 53.4 | 46.6
  Blinded reader 1 (n=93/133) | 51.9 | 51.1
  Blinded reader 2 (n=93/133) | 54.1 | 39.1
  Blinded reader 3 (n=93/133) | 52.6 | 50.4
  Clinical investigators (n=113/140) | 69.3 | 50.0
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Majority reader; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 6.8, 95% CI 2-sided [lower limit -2.2] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 1; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 0.0, 95% CI 2-sided [lower limit -9.7] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 2; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 14.3, 95% CI 2-sided [lower limit 5.1] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 3; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 3.0, 95% CI 2-sided [lower limit -5.8] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Clinical investigator; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 20.0, 95% CI 2-sided [lower limit 11.7] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

3. Primary Outcome: Specificity for Exclusion of Clinically Significant Disease Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Clinically significant disease (stenosis) was defined as 50 to 99 percent (%) stenosis of a segment, but not occluded as assessed by the SoR. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. Specificity = percentage of participants for which the imaging modalities (unenhanced or gadobutrol-enhanced) in the detection and exclusion of clinically significant stenosis.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of specificity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
Number analyzed (segments) | 1605 | 1605
percentage of specificity
  Majority reader (n=292/1605) | 94.8 | 85.7
  Blinded reader 1 (n=292/1605) | 94.4 | 83.1
  Blinded reader 2 (n=292/1605) | 94.8 | 85.0
  Blinded reader 3 (n=292/1605) | 94.0 | 80.7
  Clinical investigators (n=292/1598) | 96.5 | 83.5
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Majority reader; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 9.0, 95% CI 2-sided [lower limit 7.0] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 1; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 11.3, 95% CI 2-sided [lower limit 9.1] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 2; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 9.7, 95% CI 2-sided [lower limit 7.6] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 3; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 13.4, 95% CI 2-sided [lower limit 11.2] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Clinical investigator; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 13.1, 95% CI 2-sided [lower limit 11.0] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

4. Primary Outcome: Minimum Gadobutrol Performance for Sensitivity: Sensitivity More Than (>) 50%
Description: Clinically significant disease was defined as >50% stenosis of a segment, but not occluded as assessed by the SoR. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. Gadobutrol minimum performance criteria was based on a stenosis of 50% calculated from the native vessel diameter.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of sensitivity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA
Number analyzed (Participants) | 108
Number analyzed (segments) | 129
percentage of sensitivity
  Majority reader (n=84/119) | 54.6
  Blinded reader 1 (n=91/128) | 51.6
  Blinded reader 2 (n=82/114) | 54.4
  Blinded reader 3 (n=83/118) | 53.4
  Clinical investigators (n=108/129) | 71.3
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA; Majority reader; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 54.6, 95% CI 1-sided [lower limit 46.2]
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 1; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 51.6, 95% CI 1-sided [lower limit 43.6]
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 2; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 54.4, 95% CI 1-sided [lower limit 45.5]
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 3; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 53.4, 95% CI 1-sided [lower limit 44.8]
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA; Clinical investigator; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 71.3, 95% CI 1-sided [lower limit 64.7]

5. Primary Outcome: Minimum Gadobutrol Performance for Specificity: Specificity > 50%
Description: Clinically significant disease (stenosis) was defined as >50% stenosis of a segment, but not occluded as assessed by the SoR. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. Gadobutrol minimum performance criteria was based on a stenosis of 50% calculated from the native vessel diameter.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of specificity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA
Number analyzed (Participants) | 292
Number analyzed (segments) | 1585
percentage of specificity
  Majority reader (n=291/1555) | 95.9
  Blinded reader 1 (n=292/1585) | 95.0
  Blinded reader 2 (n=291/1554) | 96.2
  Blinded reader 3 (n=290/1544) | 95.8
  Clinical investigators (n=289/1535) | 98.4
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA; Majority reader; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 95.9, 95% CI 1-sided [lower limit 94.9]
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 1; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 95.0, 95% CI 1-sided [lower limit 93.8]
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 2; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 96.2, 95% CI 1-sided [lower limit 95.2]
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 3; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 95.8, 95% CI 1-sided [lower limit 94.8]
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA; Clinical investigator; Test type: Superiority or Other; One sided 95% confidence interval; percentage = 98.4, 95% CI 1-sided [lower limit 97.8]

6. Secondary Outcome: Length of the Right and Left Renal Arteries Assessed by Gadobutrol-enhanced MRA and Unenhanced MRA - Blinded Reader
Description: The length of the left and right renal arteries were measured from the origin at the aorta to the bifurcation into the upper and lower pole arteries or the most distal point of the renal artery which could be visualized. This distal margin was the point where the diameter was still assessable. If there were more than 2 distal branches then the first large branch that was the dominant supply to a renal pole was used as the distal point.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS
Measure: Mean (Standard Deviation); unit: millimeter(s) (mm)
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
millimeter(s) (mm)
  Left renal artery- Blind reader 1 | 35.07 (11.76) | 32.25 (11.32)
  Right renal artery - Blind reader 1 | 46.23 (14.01) | 43.05 (14.34)
  Left renal artery- Blind reader 2 | 35.07 (11.76) | 32.15 (11.35)
  Right renal artery - Blind reader 2 | 46.27 (14.01) | 42.95 (14.42)
  Left renal artery- Blind reader 3 | 35.07 (11.76) | 32.64 (12.74)
  Right renal artery - Blind reader 3 | 46.23 (14.00) | 43.05 (14.34)

7. Secondary Outcome: Length of the Right and Left Renal Arteries Assessed by Computed Tomographic Angiography (CTA) - Blinded Reader
Description: as for outcome 6
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS
Measure: Mean (Standard Deviation); unit: millimeter(s) (mm)
Arm/Group | Computed Tomographic Angiography (CTA)
Number analyzed (Participants) | 292
millimeter(s) (mm)
  Left renal artery- CTA Blind reader 4 | 36.59 (12.14)
  Right renal artery - CTA Blind reader 4 | 48.44 (14.51)
  Left renal artery- CTA Blind reader 5 | 36.59 (12.14)
  Right renal artery - CTA Blind reader 5 | 48.44 (14.50)
  Left renal artery- CTA Blind reader 6 | 36.59 (12.14)
  Right renal artery - CTA Blind reader 6 | 48.45 (14.50)

8. Secondary Outcome: Vessel Diameter (Millimeter [mm]) at the Normal Point and the Narrowest Point in Gadobutrol-Enhanced MRA, Unenhanced MRA and CTA Images
Description: The segment reduction in diameter (DIA) of greater than 10% was considered abnormal and measured. The diameter of each of these abnormal segments was measured using electronic calipers (perpendicular to the long axis of the vessel) at the point of most severe stenosis within each segment. Mean of vessel diameters was calculated by segment separately for CTA and MRA readers. For the ease of expression, the following abbreviations will be used: Diameter (DIA), Blinded Reader (BR).
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: segments
Arm/Group | Gadobutrol-Enhanced MRA | Unenhanced MRA | Computed Tomographic Angiography
Number analyzed (Participants) | 188 | 217 | 258
Number analyzed (segments) | 418 | 498 | 814
mm
  Vessel DIA at normal point: BRs | 5.13 (0.91) | 4.83 (1.05) | 5.08 (1.22)
  Vessel DIA at narrowest point: BRs | 2.80 (1.08) | 2.30 (0.99) | 2.80 (1.04)
Statistical Analysis 1: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA Minus Unenhanced MRA for blinded Reader on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.17, Standard Deviation 1.28
Statistical Analysis 2: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-Enhanced MRA for blinded reader on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = -0.09, Standard Deviation 1.14
Statistical Analysis 3: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA minus Unenhanced MRA for blinded reader on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Mean Difference = 0.41, Standard Deviation 1.15
Statistical Analysis 4: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-Enhanced MRA for blinded reader on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Diameter difference = -0.15, Standard Deviation 1.01

9. Secondary Outcome: The Percentage of Location of Stenosis >= 50% (Within and Beyond 5 Millimeter From the Aorta) in the Proximal Segments Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Location within the right and left proximal segment was based on the point of greatest stenosis and was recorded for stenosis >=50% as: - Within 5 mm of the aorta (or occlusion proximal to the origin of the segment); - Beyond 5 mm from the aorta.
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS that were evaluable; in below table, "n" signifies the number of segments that were evaluable in specified category.
Measure: Number; unit: Percentage of location
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
Percentage of location
  Within 5 mm of the aorta BR 1 (n=110; 105) | 26.4 | 22.9
  Within 5 mm of the aorta BR 2(n=83; 39) | 73.5 | 71.8
  Within 5 mm of the aorta BR 3 (n=83; 87) | 25.3 | 21.8
  Beyond 5 mm from the aorta BR 1 (n=110; 105) | 73.6 | 77.1
  Beyond 5 mm from the aorta BR 2 (n=83; 39) | 26.5 | 28.2
  Beyond 5 mm from the aorta BR 3 (n=83; 87) | 74.7 | 78.2

10. Secondary Outcome: The Percentage of Segments With Artifacts Presence
Description: Artifacts were collected for the MRA images on a segmental basis.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS
Measure: Number; unit: percentage of segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of segments
  Blinded Reader 1 | 24.7 | 92.3
  Blinded Reader 2 | 22.1 | 80.4
  Blinded Reader 3 | 41.5 | 97.4

11. Secondary Outcome: Types of Artifacts Assessed by Gadobutrol-enhanced MRA and Unenhanced MRA by Blinded Reader 1
Description: The following types of artifacts were considered: Motion artifact (including pulsatility, breathing, swallowing), venous opacification, saturation artifact (for example [eg], in-plane flow, turbulence, dephasing, saturation band), susceptibility artifacts (including devices, eg, stents), ringing artifact (eg, bands), bolus timing error, and other (artifact not specified above or no artifact).
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifact presence.
Measure: Number; unit: percentage of segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of segments
  Motion artifact | 17.5 | 81.4
  Venous opacification | 4.8 | 15.1
  Saturation artifact | 0.2 | 0.4
  Susceptibility artifacts | 0.0 | 0.1
  Other | 5.0 | 7.2

12. Secondary Outcome: Types of Artifacts Assessed by Gadobutrol-enhanced MRA and Unenhanced MRA by Blinded Reader 2
Description: as for outcome 11
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifacts presence.
Measure: Number; unit: percentage of segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of segments
  Motion artifact | 5.4 | 57.1
  Venous opacification | 12.0 | 9.6
  Saturation artifact | 0.2 | 24.4
  Susceptibility artifacts | 3.6 | 6.0
  Ringing artifact | 0.6 | 1.4
  Bolus timing error | 1.7 | 0.1
  Other | 1.7 | 6.5

13. Secondary Outcome: Types of Artifacts Assessed by Gadobutrol-enhanced MRA and Unenhanced MRA by Blinded Reader 3
Description: as for outcome 11
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifacts presence.
Measure: Number; unit: percentage of segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of segments
  Motion artifact | 32.8 | 96.2
  Venous opacification | 14.2 | 34.5
  Saturation artifact | 3.0 | 56.0
  Susceptibility artifacts | 4.0 | 7.0
  Ringing artifact | 6.7 | 76.7
  Bolus timing error | 0.3 | 1.5
  Other | 0.7 | 0.2

14. Secondary Outcome: The Percentage of Accessory (Non-dominant) Renal Artery Presence Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: An accessory renal artery was defined as an additional, non-dominant, renal artery typically emanating from the aorta and anastomosing distal to the proximal third, segment of that renal artery. It was recorded only as present or absent on the right and left, regardless of how many accessory renal arteries were present.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of accessory
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of accessory
  Left side: Reader 1 | 7.2 | 0.7
  Right side: Reader 1 | 9.2 | 1.4
  Left side: Reader 2 | 15.4 | 2.7
  Right side: Reader 2 | 17.8 | 3.1
  Left side: Reader 3 | 13.4 | 5.8
  Right side: Reader 3 | 16.4 | 4.5
  Left side: Clinical investigators | 18.2 | 11.6
  Right side: Clinical investigators | 19.2 | 12.7

15. Secondary Outcome: The Presence of Any Aneurysmal Dilatation in Each Segment (Proximal, Mid- and Distal) in the Right and the Left Renal Arteries Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Any focal dilatation (aneurysmal dilatation) of a segment was recorded. The diameter at the widest point was measured with the electronic calipers if a dilatation was present in any segment. The number of participants with an aneurysmal dilatation in each segment (proximal, mid- and distal) in the right and the left renal arteries assessed by gadobutrol-enhanced MRA and unenhanced MRA were reported.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of participants
  Right : Proximal | 0.3 | 0
  Right : Mid | 1.0 | 0
  Right : Distal | 1.4 | 0
  Left : Proximal | 0 | 0
  Left : Mid | 0.3 | 0.3
  Left : Distal | 0.7 | 0.3

16. Secondary Outcome: The Percentage of Participants With Diagnosis of Fibromuscular Dysplasia and Arteriosclerosis Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: as for outcome 15
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of participants
  Fibromuscular dysplasia : reader 1 | 2.7 | 0.7
  Arteriosclerotic : reader 1 | 16.4 | 12.0
  Fibromuscular dysplasia : reader 2 | 4.1 | 0.0
  Arteriosclerotic : reader 2 | 38.4 | 18.8
  Fibromuscular dysplasia : reader 3 | 6.2 | 0.7
  Arteriosclerotic : reader 3 | 41.1 | 54.5

17. Secondary Outcome: Diagnostic Confidence by the Blinded Readers Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Diagnostic confidence was evaluated to determine the level of certainty that the blinded readers assigned to a diagnosis for each segment. This was defined as the degree of confidence that the information on the MRA images represented the true and complete clinical picture of a particular segment. The degree of confidence was rated on a 4-point scale: 1=Not confident; 2=Somewhat confident; 3=Confident; 4=Very confident.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; In the below table, "n" signifies the number of segments that were evaluable in specified category.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 291
Units on scale
  Blinded reader 1(n=1745; 1728) | 3.0 (0.8) | 1.9 (0.7)
  Blinded reader 2 (n=1745; 1729) | 3.5 (0.8) | 2.1 (1.0)
  Blinded reader 3 (n=1749; 1737) | 3.5 (0.8) | 2.2 (0.9)

18. Secondary Outcome: The Percentage of Participants With Additional Imaging Studies Recommended by the Blinded Readers and the Clinical Investigator After Evaluation of the Gadobutrol-Enhanced and Unenhanced MRA Images
Description: A measure of diagnostic value was the reduction in the number of additional diagnostic imaging studies recommended/ordered. The clinical investigators and the blinded readers were asked if they had recommended an additional imaging study for each participant, and the data were recorded.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 292 | 292
percentage of participants
  Blinded reader 1 | 41.4 (0.8) | 96.6 (0.7)
  Blinded reader 2 | 14.0 (0.8) | 77.1 (1.0)
  Blinded reader 3 | 8.6 (0.8) | 44.9 (0.9)
  Clinical investigators | 18.8 | 43.5

19. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Gadobutrol-Enhanced and Unenhanced MRA Images - Blinded Reader 1
Description: An additional imaging study recommended was specified from the following list: Non-contrast MRA, Contrast-enhanced MRA, CTA, Ultrasound, Digital subtraction catheter angiogram (DSCA), and Nuclear medicine study.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS with participants who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 121 | 282
participants
  Non-contrast MRA | 0 (0.8) | 2 (0.7)
  Contrast-enhanced MRA | 1 (0.8) | 0 (1.0)
  CTA | 120 (0.8) | 280 (0.9)
  Ultrasound | 0 | 0
  DSCA | 0 | 0
  Nuclear medicine study | 0 | 0

20. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Gadobutrol-Enhanced and Unenhanced MRA Images - Blinded Reader 2
Description: as for outcome 19
Time Frame: Images were taken pre-injection and post-injection
Population: FAS with participants who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 41 | 225
participants
  Non-contrast MRA | 0 (0.8) | 0 (0.7)
  Contrast-enhanced MRA | 0 (0.8) | 114 (1.0)
  CTA | 39 (0.8) | 110 (0.9)
  Ultrasound | 1 | 1
  DSCA | 1 | 0
  Nuclear medicine study | 0 | 0

21. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Gadobutrol-Enhanced and Unenhanced MRA Images - Blinded Reader 3
Description: as for outcome 19
Time Frame: Images were taken pre-injection and post-injection
Population: FAS with participants who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 25 | 131
participants
  Non-contrast MRA | 0 (0.8) | 1 (0.7)
  Contrast-enhanced MRA | 1 (0.8) | 14 (1.0)
  CTA | 22 (0.8) | 116 (0.9)
  Ultrasound | 0 | 0
  DSCA | 2 | 0
  Nuclear medicine study | 0 | 0

22. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Clinical Investigator After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images
Description: as for outcome 19
Time Frame: Images were taken pre-injection and post-injection
Population: FAS with participants who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 55 | 127
participants
  Non-contrast MRA | 0 (0.8) | 0 (0.7)
  Contrast-enhanced MRA | 2 (0.8) | 114 (1.0)
  CTA | 50 (0.8) | 12 (0.9)
  Ultrasound | 0 | 0
  DSCA | 3 | 1
  Nuclear medicine study | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were assessed from the time the consent was signed until 72 (±6) hours follow-up after the study MRA and continued until the end of the study (either the 72 hour follow-up or the CTA, if performed after the MRA as part of the study).
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Serious Adverse Events (participants affected / at risk) | 0/315
Other Adverse Events (participants affected / at risk) | 14/315
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol (Gadavist, BAY 86-4875) (N=315)
Nausea (Gastrointestinal disorders) | 8
Headache (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other